CLINICAL TRIAL: NCT00411359
Title: Cardiac Rehabilitation for the Treatment of Refractory Angina
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart and Lung Institute (Other)
Collaborators: British Heart Foundation (Other); Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Prof. Peter Collins, Professor of Clinical Cardiology, National Heart and Lung Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06/Q0404/77; PG/06/087/21239 (Other Grant/Funding Number: British Heart Foundation)
Record Dates: First submitted 2006-12-12; First posted 2006-12-14 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Angina Pectoris; Coronary Disease
Keywords: Refractory angina; Cardiac rehabilitation; Symptomology; Physical ability; Exercise; Psychology; Quality of life; Risk factors
MeSH Terms: conditions — Angina Pectoris; Coronary Disease; Motor Activity | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cardiac rehabilitation (Experimental): 8-week cardiac rehabilitation programme
  Interventions: Behavioral: Cardiac rehabilitation
- Monitoring (No Intervention): Carry on life as normal

INTERVENTIONS:
Behavioral: Cardiac rehabilitation — Phase III cardiac rehabilitation programme
  Arms: Cardiac rehabilitation

SUMMARY:
The purpose of this study is to determine whether cardiac rehabilitation is a successful treatment for refractory angina, in relation to improvements in cardiovascular risk factors, physical ability, symptomology, quality of life and psychological morbidity.

DETAILED DESCRIPTION:
The majority of patients presenting with angina pectoris resulting from coronary artery disease (CHD) are successfully treated with interventions including coronary artery bypass grafting (CABG) and percutaneous transluminal coronary angioplasty (PTCA) and medical management. However, a growing number of patients experience persistent angina in spite of intervention and optimal medical treatment. Such patients are referred to as suffering from 'refractory angina'.

Currently, cardiac rehabilitation centres are reluctant to accept patients with ongoing angina or complicated cardiovascular history, in spite of the duration or stability of the symptoms. Indeed, angina and heart failure are often used to exclude patients from cardiac rehabilitation. However, in the recent updated American Heart Association (AHA) recommendations for exercise and training, cardiac rehabilitation and supervised exercise training is recommended for patients with ongoing angina, previous history of CABG, MI, PTCA and patients with existing cardiomyopathy in order to promote a reduction in myocardial ischaemia at rest and during sub-maximal exercise, while reducing the risk for the progression of CHD. Nevertheless, studies exploring the physiological and psychological impact of routinely available CR as a stand-alone intervention among refractory angina patients have not previously been undertaken. Until such studies are performed, CR practitioners will continue to refuse to accept refractory angina patients for participation in CR.

Research questions:

* Is an eight-week cardiac rehabilitation exercise programme an appropriate treatment option for patients with refractory angina?
* Does an eight-week cardiac rehabilitation exercise programme improve the physical functioning and cardiovascular health of patients with refractory angina?
* Is symptom severity and frequency reduced following an eight-week cardiac rehabilitation exercise programme in patients with refractory angina?
* Does an eight-week cardiac rehabilitation exercise programme have any impact on anxiety, depression, cardiac anxiety and quality of life in patients with refractory angina?
* Are any physiological or psychological effects acquired by patients with refractory angina participating in a cardiac rehabilitation exercise programme maintained at an eight-week follow-up?

The study is conceived as a randomised intervention-control study of a standard, routinely available Phase III hospital-based CR program among patients with refractory angina. Patients will be randomly assigned to an eight-week CR programme based at Harefield Hospital or symptom diary monitoring control group.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with refractory angina > 6 months
* Two or more episodes of angina per week
* Males and females aged 30 - 80
* Previous history of single or multiple myocardial infarction (MI), coronary artery bypass graft (CABG), percutaneous transluminal coronary angioplasty (PTCA) or any combination of the above
* Prescribed optimal medical therapy
* AHA exercise and training guidelines classification B and C
* Willing to give written informed consent

Exclusion Criteria:

* History of any other chronic illness
* AHA exercise and training guidelines classification class D
* Suffer any physical condition for which exercise is a contra-indication
* Participation in two or more periods of planned moderate intensity exercise per week during the past 6 months
* Participation in another research study within the previous 60 days
* History of psychiatric illness
* Unwilling to give written informed consent

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2006-12; Primary Completion 2009-12 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Health anxiety | Base, week 8 (post intervention/monitoring), week 16 (8 weeks post intervention/monitoring)
  Health anxiety questionnaire (HAQ)
Generalised anxiety and depression | Base, week 8 (post intervention/monitoring), week 16 (8 weeks post intervention/monitoring)
  Hospital Anxiety and Depression scale (HADS)

SECONDARY OUTCOMES:
Systolic and diastolic blood pressure | Base, week 8 (post intervention/monitoring), week 16 (8 weeks post intervention/monitoring)
  Measured after 10 minutes sitting, using automated machine (eg. Omron machine)
Heart rate | Base, week 8 (post intervention/monitoring), week 16 (8 weeks post intervention/monitoring)
  Heart rate measured using automated machine (eg. Omron blood pressure machine) or manually at the radial pulse
Anthropomometry | Base, week 8 (post intervention/monitoring), week 16 (8 weeks post intervention/monitoring)
  Weight, height, waist circumference (tape measure), hip circumference (tape measure), body mass index calculated from height and weight using the following website: http://www.nhlbisupport.com/bmi/bmi-m.htm
Fasting lipids | Base, week 8 (post intervention/monitoring), week 16 (8 weeks post intervention/monitoring)
  total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides. Measured in biochemistry departments of the Royal Brompton & Harefield NHS Foundation Trust using standard techniques.
Social support | Baseline
  Measured using the ENRICHED social support instrument (ESSI)
Angina related health beliefs | Base, week 8 (post intervention/monitoring), week 16 (8 weeks post intervention/monitoring)
  Measured using the York angina beliefs scale.
Physical activity and exercise capacity | Base, week 8 (post intervention/monitoring), week 16 (8 weeks post intervention/monitoring)
  Progressive shuttle walk test
Angina frequency and severity | Base, week 8 (post intervention/monitoring), week 16 (8 weeks post intervention/monitoring)
  Subjects completed a daily symptom monitoring diary
Quality of life | Base, week 8 (post intervention/monitoring), week 16 (8 weeks post intervention/monitoring)
  SF-36 quality of life scale
Plasma glucose | Base, post intervention/monitoring, 8 weeks post intervention/monitoring
  Measured in the biochemistry departments of the Royal Brompton & Harefield NHS Foundation Trust using standard techniques.
Urea & electrolytes | Base, post intervention/monitoring, 8 weeks post intervention/monitoring
  Measured in the biochemistry departments of the Royal Brompton & Harefield NHS Foundation Trust using standard techniques
Liver function tests | Baseline, post intervention/monitoring, 8 weeks post intervention/monitoring
  Measured in the biochemistry departments of the Royal Brompton & Harefield NHS Foundation Trust using standard techniques.
Thyroid function tests | Baseline, post intervention/monitoring, 8 weeks post intervention/monitoring
  Measured in the biochemistry departments of the Royal Brompton & Harefield NHS Foundation Trust using standard techniques.
Hb | Baseline, post intervention/monitoring, 8 weeks post intervention/monitoring
  Measured in the haematology departments of the Royal Brompton & Harefield NHS Foundation Trust using standard techniques.
HbA1C (if diabetic) | Baseline, post intervention/monitoring, 8 weeks post intervention/monitoring
  Measured in the haematology department of the Royal Brompton & Harefield NHS Foundation Trust using standard techniques

CONTACTS AND LOCATIONS:
Overall Officials: Peter Collins, MA, MD, FRCP, Principal Investigator — National Heart and Lung Institute, Imperial College London; Kim Fox, MD, FRCP, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust; Mahmud Barbir, FRCP, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- National Heart and Lung Institute, Imperial College London, London, United Kingdom

REFERENCES:
- [Background] Mannheimer C, Camici P, Chester MR, Collins A, DeJongste M, Eliasson T, Follath F, Hellemans I, Herlitz J, Luscher T, Pasic M, Thelle D. The problem of chronic refractory angina; report from the ESC Joint Study Group on the Treatment of Refractory Angina. Eur Heart J. 2002 Mar;23(5):355-70. doi: 10.1053/euhj.2001.2706. No abstract available. PMID 11846493
- [Background] DeJongste MJ, Tio RA, Foreman RD. Chronic therapeutically refractory angina pectoris. Heart. 2004 Feb;90(2):225-30. doi: 10.1136/hrt.2003.025031. No abstract available. PMID 14729809
- [Background] Gowda RM, Khan IA, Punukollu G, Vasavada BC, Nair CK. Treatment of refractory angina pectoris. Int J Cardiol. 2005 May 11;101(1):1-7. doi: 10.1016/j.ijcard.2004.03.066. PMID 15860376
- [Background] Chester M, Hammond C, Leach A. Long-term benefits of stellate ganglion block in severe chronic refractory angina. Pain. 2000 Jul;87(1):103-105. doi: 10.1016/S0304-3959(00)00270-0. PMID 10863051
- [Background] Stewart S. Refractory to medical treatment but not to nursing care: can we do more for patients with chronic angina pectoris? Eur J Cardiovasc Nurs. 2003 Sep;2(3):169-70. doi: 10.1016/S1474-5151(03)00067-7. No abstract available. PMID 14622623
- [Background] Moore RK, Groves D, Bateson S, Barlow P, Hammond C, Leach AA, Chester MR. Health related quality of life of patients with refractory angina before and one year after enrolment onto a refractory angina program. Eur J Pain. 2005 Jun;9(3):305-10. doi: 10.1016/j.ejpain.2004.07.013. PMID 15862480
- [Background] Lear SA, Ignaszewski A. Cardiac rehabilitation: a comprehensive review. Curr Control Trials Cardiovasc Med. 2001;2(5):221-232. doi: 10.1186/cvm-2-5-221. PMID 11806801
- [Background] Hevey D, Brown A, Cahill A, Newton H, Kierns M, Horgan JH. Four-week multidisciplinary cardiac rehabilitation produces similar improvements in exercise capacity and quality of life to a 10-week program. J Cardiopulm Rehabil. 2003 Jan-Feb;23(1):17-21. doi: 10.1097/00008483-200301000-00004. PMID 12576907
- [Background] Grace SL, Abbey SE, Shnek ZM, Irvine J, Franche RL, Stewart DE. Cardiac rehabilitation I: review of psychosocial factors. Gen Hosp Psychiatry. 2002 May-Jun;24(3):121-6. doi: 10.1016/s0163-8343(02)00178-0. PMID 12062135
- [Background] Grace SL, Abbey SE, Shnek ZM, Irvine J, Franche RL, Stewart DE. Cardiac rehabilitation II: referral and participation. Gen Hosp Psychiatry. 2002 May-Jun;24(3):127-34. doi: 10.1016/s0163-8343(02)00179-2. PMID 12062136
- [Background] Johnston M, Foulkes J, Johnston DW, Pollard B, Gudmundsdottir H. Impact on patients and partners of inpatient and extended cardiac counseling and rehabilitation: a controlled trial. Psychosom Med. 1999 Mar-Apr;61(2):225-33. doi: 10.1097/00006842-199903000-00015. PMID 10204976
- [Background] Yoshida T, Kohzuki M, Yoshida K, Hiwatari M, Kamimoto M, Yamamoto C, Meguro S, Endo N, Kato A, Kanazawa M, Sato T. Physical and psychological improvements after phase II cardiac rehabilitation in patients with myocardial infarction. Nurs Health Sci. 1999 Sep;1(3):163-70. doi: 10.1046/j.1442-2018.1999.00021.x. PMID 10894639
- [Background] Fletcher GF, Balady GJ, Amsterdam EA, Chaitman B, Eckel R, Fleg J, Froelicher VF, Leon AS, Pina IL, Rodney R, Simons-Morton DA, Williams MA, Bazzarre T. Exercise standards for testing and training: a statement for healthcare professionals from the American Heart Association. Circulation. 2001 Oct 2;104(14):1694-740. doi: 10.1161/hc3901.095960. No abstract available. PMID 11581152
- [Background] Taylor RS, Brown A, Ebrahim S, Jolliffe J, Noorani H, Rees K, Skidmore B, Stone JA, Thompson DR, Oldridge N. Exercise-based rehabilitation for patients with coronary heart disease: systematic review and meta-analysis of randomized controlled trials. Am J Med. 2004 May 15;116(10):682-92. doi: 10.1016/j.amjmed.2004.01.009. PMID 15121495
- [Background] Asbury EA, Creed F, Collins P. Distinct psychosocial differences between women with coronary heart disease and cardiac syndrome X. Eur Heart J. 2004 Oct;25(19):1695-701. doi: 10.1016/j.ehj.2004.07.035. PMID 15451147
- [Result] Asbury EA, Webb CM, Probert H, Wright C, Barbir M, Fox K, Collins P. Cardiac rehabilitation to improve physical functioning in refractory angina: a pilot study. Cardiology. 2012;122(3):170-7. doi: 10.1159/000339224. Epub 2012 Jul 27. PMID 22846707